CLINICAL TRIAL: NCT03732755
Title: An Open-label Study of Safety and Effectiveness of the Portable Neuromodulation Stimulator (PoNS®) Treatment for Subjects With a Chronic Balance Deficit Due to Mild-to-moderate Traumatic Brain Injury (TBI)
Brief Title: PoNS Clinical Experience Program (TBI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Helius Medical Inc (Industry)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHC-TBI-PoNS-CE KESSLER
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Mild to Moderate Traumatic Brain Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active (Experimental): PoNS Treatment will consist of three stages: an in-clinic training program, a home training program, and an extended home training program. During all stages of the study, subjects will complete three training sessions per day, morning, afternoon and evening, 6 days per week.
  Interventions: Device: PoNS Treatment

INTERVENTIONS:
Device: PoNS Treatment — PoNS Treatment will consist of three stages: an in-clinic training program, a home training program, and an extended home training program. During all stages of the study, subjects will complete three training sessions per day, morning, afternoon and evening, 6 days per week.
  Daily Training Program: The same daily training program will be performed during all stages with the exception of the morning BAT session, which is not performed during stage 2 or 3:
  Morning:
  Warm Up Exercises without the PoNS Balance Training with PoNS Gait Training with PoNS Breathing and Awareness Training (BAT) with PoNS 3- to 4-hour break between morning and afternoon sessions
  Afternoon:
  Balance Training with PoNS Movement Control Training without PoNS Gait Training with PoNS
  Evening:
  Breathing and Awareness Training with PoNS To be performed at home during all stages

SUMMARY:
- Brief Summary: Prospective, cohort, open-label study. The cohort consists of people who have a chronic balance dysfunction due to a mild to moderate traumatic brain injury (TBI). All participants will participate in a 14-week PoNS Treatment protocol - a combination of symptom specific physical exercises and repeated use of the PoNS device.

Subjects who meet the initial screening entrance criteria will be scheduled for a baseline assessment to evaluate balance and gait. Subjects will then begin the PoNS Treatment program and re-perform some assessments at 2, 5 and 14 weeks evaluating their functional improvements.

ELIGIBILITY:
Inclusion Criteria:

- 1. At least 18 years of age, inclusive, at the time of screening. 2. Acceptable results (as determined by the investigator) of a full history and physical performed or supervised by the investigator at each site. This will include a careful examination of the tongue and oral cavity for any abnormalities. History should include the nature and duration of any prior physical therapy program the subject may have participated in to address the balance and/or gait symptoms of their TBI.

3. Documentation on the history of a qualifying TBI, mild to moderate in severity. For reference, the Armed Forces Health Surveillance Branch (AFHSB) definitions of mild and moderate TBI will be used. The definitions are as follows:

* Mild TBI: Confused or disoriented state which lasts less than 24 hours; or loss of consciousness for up to 30 minutes, or memory loss lasting less than 24 hours. Excludes penetrating TBI.
* Moderate TBI: Confused or disoriented state which lasts more than 24 hours; and/or loss of consciousness for more than 30 minutes but less than 24 hours, or memory loss lasting greater than 24 hours but less than seven days; or meets criteria for Mild TBI except an abnormal CT scan is present. Excludes penetrating TBI.

The investigator will ascertain whether the prior medical records are sufficiently detailed to support the classification of the TBI.

4. Acceptable results from within the last three (3) months as determined by the site investigator of basic standard blood work to include CBC, TSH, HbA1C, Liver and Kidney panels, and a 12-lead ECG with automated reporting capability. Any abnormal result that is judged clinically significant by the investigator will be communicated to the subject and if treated by their personal physician and deemed recovered, the subjects may be reconsidered for inclusion. If the investigator is uncertain he or she will communicate with the Sponsor's Medical Officer.

5. If female, the subject is not pregnant, not breastfeeding and has a negative pregnancy test prior to receipt of the PoNS device

- Note: Pregnancy testing will be repeated at end-of-study (EOS) (i.e., end of at- home period).

6. If female is of childbearing potential, the subject agrees to use adequate contraception from screening and throughout the study period.

A female of non-childbearing potential is defined as a subject who is postmenopausal (continuous amenorrhea for 12 months) or surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

7. Balance disorder as indicated by the NeuroCom® Sensory Organization Test (SOT) composite score at least 16 points below normal [adjusted for age and height, based on normative data] due to a mild-to-moderate traumatic brain injury (TBI).

8. At least three (3) months post most recent TBI at the time of screening. 9. Stable neurologic status, as determined from subject's medical records and the study physician's opinion based on no new or changing symptoms.

10. Qualifying MRI report to be entered into the data collection form. For all participants who do not have a qualifying MRI, a new MRI will be obtained.

11. Ambulatory and able to walk continuously over-ground or on a treadmill for 20 minutes, level grade (no inclination) and at any speed, with support, if needed.

12. Able to understand the study procedures and give informed consent. 13. Willing and able to adhere to the study schedule. 14. Willing to complete a neuropsychological evaluation if deemed necessary by the investigator prior to inclusion in the study.

Exclusion Criteria:

1. Medical findings from screening history, physical examination or radiological test that the investigator deems clinically significant or that would otherwise impact patient safety or data integrity.
2. Planned use or use of any investigational product (i.e., not approved by the FDA), pharmaceutical or device, within 30 days preceding receipt of the PoNS device and during the entire period of subject participation.
3. Any previous use of the Portable Neuromodulation Stimulator (PoNS)
4. Balance or gait deficits due to lower extremity injury or neurological condition other than TBI.
5. Severe TBI defined as an injury with a confused or disoriented state which lasts more than 24 hours; and/or loss of consciousness for more than 24 hours, or memory loss for more than seven days.
6. Penetrating brain injury, refractory subdural hematoma, or craniotomy unrelated to the resolution of qualifying traumatic brain injury. Investigator discretion may be exercised on an individual case where surgery was performed that did not remove or significantly alter brain tissue (e.g., to treat a brain aneurysm). Surgery must have been performed at least 6 months prior to screening and a CT scan must be provided to demonstrate no large residual lesions.
7. Oral health problems active at the time of recruitment. Any history of oral health problems (e.g., gum disease or cankers) will be noted on the data collection form.
8. Oral surgery within 3 months of screening.
9. History of oral cancer.
10. Non-removable metal orthodontic devices (e.g., braces) or oral cavity piercings that could interfere with PoNS use.
11. Presence of metallic implant or other MRI-incompatible device.
12. Known allergy to gold, nickel or copper.
13. Blood pressure abnormalities considered clinically significant by the study physician. If the subject has a systolic blood pressure of <100 mmHg, they will be evaluated for orthostatic hypotension and if the investigator deems this a risk for the subject's health or safety they will be excluded. If systolic blood pressure >160 mm Hg (average of 3 measurements) at screening and the subject is on medications, the subject will be referred back to their family doctor for review and control but can be re-evaluated once the treating physician deems them to have stable blood pressure.

    - Note: BP should be measured seated, legs uncrossed, after resting for 5 minutes, with measurements taken 2 minutes apart. Two BP readings should be taken and averaged. If the first two readings differ by >5 mm Hg, a third measurement should be taken and an average calculated for all 3 values.
14. Use of Coumadin or any other anticoagulant other than aspirin in the last six months.
15. Untreated or undiagnosed diabetes - the subject will be referred to their family physician and may be re-evaluated at a later date. Undiagnosed diabetes is defined as an HbA1C taken during screening above the upper limit of normal at the study site.
16. Diabetic neuropathy.
17. Active or recent (within 1 year) treatment for any cancer, excluding basal cell carcinoma.
18. Neurological disorders other than those attributed to the primary diagnosis, (e.g., neurodegenerative diseases such as Multiple Sclerosis (MS), Parkinson's disease (PD), Alzheimer's disease (AD) or other dementia, Amyotrophic Lateral Sclerosis (ALS). Lower back pain, lumbar spine abnormalities, or history of lumbar spine surgery with no residual clinical significant lower extremity weakness are not excluded.
19. History of epileptic or other seizure disorders .
20. Known ischemic heart disease (angina, stent, history of myocardial infarction, >70% stenosis or cardiovascular imaging) and/or history or atrial or ventricular arrhythmias with or without syncope. Any abnormality on the screening ECG will be referred to the subject's family physician for evaluation and clearance and then the subject can be re-evaluated for inclusion in the study.
21. Any other untreated or unstable acute or chronic, clinically significant medical condition for which the subject is currently undergoing treatment (e.g., autoimmune or immunodeficient disorders) and that the investigator deems unsuitable for inclusion.
22. Use of a lower extremity biomechanical prosthetic with the exception of a splint to address foot drop.
23. Chronic use of any potentially interfering drug such as a neuroactive (ototoxic, anti-seizure, anti-convulsive) medication, or chronic/PRN use of any medication that would, in the opinion of the investigator, compromise the subject's ability to function or perform the study activities.
24. Addition of and/or major change in type or dosage of any prescription medication within 3 months prior to receipt of the PoNS device at the time of screening, subject to physician discretion.
25. Active alcoholism documented by the investigator at the time of screening. The investigator will have the right to exclude subject participation if, in their opinion, the subject seems intoxicated at time of screening and/or during any study appointment.
26. History of drug abuse as documented by the investigator at the time of screening. The investigator will have the right to exclude subject participation if, in their opinion, the subject seems intoxicated at time of screening or presentation for treatment
27. Recent (6 months) history of smokeless tobacco use (i.e., chewing tobacco, oral tobacco, spit or spitting tobacco, dip, chew, snuff*) (*NCI definition)

    a. Note: Cigarette, cigar, pipe, and/or e-cigarette use is not exclusionary
28. Any reason, considered by the principal investigator or designee to preclude subject enrollment in the study that might represent a threat to health, safety, or an inability to comply with the study protocol.
29. Subject is incompatible with the device.
30. Subject is currently in a focused physical rehabilitation program for balance or gait symptoms resulting from their TBI and has not been deemed by their treating clinician to have reached a plateau.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in balance score (SOT) from baseline to the end of 14 weeks | Baseline, 2 weeks, 5 weeks and 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Institute for Rehabilitation and Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No